CLINICAL TRIAL: NCT06042803
Title: Clinical Lactation Study on the Exposure to Medicines Via Human Milk: an Umbrella Study Protocol
Brief Title: UmbrelLACT Study: Clinical Lactation Study on the Exposure to Medicines Via Human Milk
Acronym: UmbrelLACT
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Innovative Medicines Initiative (Other); BELpREG (Unknown)
Responsible Party: Sponsor
Other Study IDs: S67204
Record Dates: First submitted 2023-08-07; First posted 2023-09-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-06

CONDITIONS: Breast Feeding; Human Milk
Keywords: Infant exposure; Physiologically-based pharmacokinetic models; Neonatology; breastfeeding; Pharmacology; Medicines; Drug transfer; Medication intake
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human milk samples Optionally, plasma samples
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Human milk collection — Every time the mother would normally feed the child, we ask to collect the total milk volume for the feed from both breasts by an electric pump. For each collection, the volume and time will be noted, the container will be inverted and 5 to 10ml of that volume will be transferred in a polypropylene test tube or other tube type depending on the type of compounds (=sample to determine drug concentration in milk) for analysis (max 10% of the collected volume of each feed). The participant decides how the remainder of the collected milk is used. The milk samples will immediately be stored in the refrigerator (4°C) after being labeled. The samples will be collected by one of the investigators within 24 hours, will be transported on ice and frozen at -80°C until analysis.
Other: Optionally: maternal blood sample — Blood collection to determine the drug concentration in plasma (6 to 10mL EDTA or other tube type, depending on the type of compound) will be performed at least within 1 hour interval with the first feeding (pumping) after medication intake, and 24 hours after medication intake (with preferable milk collection within 1 hour of blood sampling). The sample label, date and time of sampling will be noted.
Other: Optionally: child blood sample — Blood collection of the infant to determine systemic exposure of child(1-5% of the total blood volume, according to the FDA guidelines, in an EDTA or other tube type, depending on the type of compound,) will be performed at the same day as the maternal sampling, if parental consent is obtained. The sample label, date and time of sampling will be noted.

SUMMARY:
The goal of this observational study is to determine the concentration of medicines in human milk during maternal medicine intake. The main questions it aims to answer are:

* What is the concentration of maternal medicines in human milk?
* What is the (estimated) intake and exposure in the breastfed infant?

Participants will be asked to

* fill out a questionnaire regarding medical data of the mother and child
* track medication intake for 3 days
* collect milk samples during 24 hours
* optionally, donate 2 blood samples of the mother and give consent to one blood sample of the child
* fill out a questionnaire regarding the general health of the child.

DETAILED DESCRIPTION:
There is an immense information gap regarding safety of medicines during lactation which can result in a lack of breastfeeding adherence. According to literature, 50% of women need pharmacotherapy in the postpartum period. However, the proportion of nursing women in need of medication rises, due to later age pregnancies and the increased prevalence of chronic diseases. Evidence-based decisions on the use and selection of medicine during breastfeeding are challenging for many medicines, due to the lack of available information, such as cardiovascular compounds (e.g. atorvastatin, simvastatin), antidepressants (e.g. venlafaxine), anti-epileptics (e.g. topiramate, pregabalin), etc. This often results in unnecessary cessation of breastfeeding or poor adherence to/avoidance of pharmacological treatment.

The objective of this prospective trial is to collect information about the human milk transfer of maternal medicines, subsequent infant exposure, and general health outcome of the infant. Furthermore, the data of this clinical lactation study will be used to verify the performance of pharmacologically-based pharmacokinetic (PBPK) models to predict disposition of medicines in human milk and subsequent neonatal exposure during lactation. An umbrella protocol approach is used. This means that each request or compound for which milk samples might be collected / offered by women, will be reviewed and evaluated for feasibility and relevance.

The investigators expect to enroll 5, at maximum 15, mothers per year, who have been prescribed maternal medication for medical reasons and are breastfeeding their infant (/expressing milk) while taking this medication. The participating mother will be asked to collect milk samples and optionally to donate 2 blood samples during 24h: one at the time of milk pumping the first time after medication intake and one at the last pumping session of the 24h period. The parents can optionally consent for collecting a blood sample of the infant for the study (1-5% of the total blood volume, according to the FDA guidelines). In addition, clinical maternal and infant variables will be collected, as well as medication regimen, sampling details and general infant health information using 2 questionnaires.

To conclude, with this study data about the concentration of maternal medication in human milk, and the exposure in the nursing infant will be generated. This information is an essential first step towards evidence-based risk assessment on the use of drugs during lactation.

ELIGIBILITY:
Inclusion Criteria:

* For breastfeeding women

  * Maternal age: ≥ 18 year
  * Currently exclusively or partially breastfeeding (/expressing milk) at the time of milk sampling
  * Using medicines for any indication, with at least 5 half-lives of the medicine taken
  * Willing to express and collect human milk
  * Signed informed consent to participate and for processing their personal data
* For infants

  * Gestational age at birth: ≥24 weeks
  * Parental signed informed consent to participate and for processing their personal data

Exclusion Criteria:

* Maternal age <18 years
* Mother of twins
* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinicians from University Hospitals Leuven and other healthcare facilities can give women who are breastfeeding or expressing milk and are actively taking maternal medicines, the contact information of the study team. Furthermore, the study background and contact information of the study team are available through the BELgPREG project (www.belpreg.be), a research initiative on the use of medicines during pregnancy. The study team will not interfere with the decision to prescribe medicines or to breastfeed. If interested, women can contact a study team member who will plan an information moment (by phone or video call) to explain the study and informed consent.
  Healthy volunteers are healthy breastfeeding women, >18 years and willing to donate a milk sample and optionally a plasma sample.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The concentration of maternal medicines in human milk | 24 hours (sampling day)
  * Quantification of the concentration of medicines in human milk: concentration, milk-to-plasma (M/P) ratio;
  * The PK parameters of medicines and relevant metabolites in human milk: area under the milk concentration-time curve (AUC), the average concentration (AUC divided by dosing interval), peak and trough milk concentrations (if available, depending on dosing regimen and lactation regimen), and time to reach peak milk concentration.
  * The PK parameters of medicines and relevant metabolites in plasma from lactating women compared to available scientific literature results, such as AUC, peak plasma concentration, time to peak plasma concentration, plasma clearance or apparent oral clearance, apparent volume of distribution and terminal half-life.

SECONDARY OUTCOMES:
The estimated intake of medicines in the nursing infant via human milk: DID | 24 hours (sampling day)
  The daily infant dosage (DID)(mg/d)
  = ∑(total drug concentration in each milk collection x expressed milk volume in each milk collection)
The estimated intake of medicines in the nursing infant via human milk: eDID - maxDID | 24 hours (sampling day)
  The estimated Daily infant dosage (eDID)(mg/kg/d) and the infant risk (maxDID) expressed as a daily weight normalized dose (mg/kg/d), with 150mL/kg/d and 200mL/kg/d as maximum estimated milk intake, respectively. The calculation of the M/P ratio is based on the AUC on multiple time points, if possible.
  = M/P ratio x average plasma concentration x estimated milk intake
The estimated intake of medicines in the nursing infant via human milk: RID | 24 hours (sampling day)
  The relative infant dose (RID)(%)
  = [eDID (mg/kg/d)/Maternal Dosage (mg/kg/d)] x 100
The estimated intake of medicines in the nursing infant via human milk: RIDtherapeutic | 24 hours (sampling day)
  The relative infant therapeutic dose (RIDtherapeutic)(%)
  = [estimated daily infant dosage (mg/kg/d)/Daily therapeutic infant dosage (mg/kg/d)] x 100
The estimated intake of medicines in the nursing infant via human milk: Css, ave | 24 hours (sampling day)
  The average infant medicine concentration at steady state (Css, ave)(ng/mL), if oral bioavailability (F) and drug clearance (CL) are known for the paediatric population
  = oral bioavailability (F) x [eDID (mg/kg/d)/Clearance (CL; L/d)]x1000
The systemic exposure to medicines in the nursing infant via breastfeeding: infant systemic medicine concentration | 24 hours (sampling day)
  The measured infant systemic medicine concentration if the parents give consent for collection of a blood sample from the infant;
The systemic exposure to medicines in the nursing infant via breastfeeding: infant/maternal plasma ratio | 24 hours (sampling day)
  The infant/maternal plasma ratio if a blood sample from the infant is available;
The systemic exposure to medicines in the nursing infant via breastfeeding | 24 hours (sampling day)
  Rate of medicine absorption in infants through human milk (e.g., infant plasma concentration/milk concentration) if a blood sample from the infant is available;
The general health status (including possible adverse effects) of the nursing infant | 2 weeks (in case of an acute maternal treatment/condition) or 2 months (in case of an chronic maternal treatment/condition)
  The general health status of the infant, reported by maternal questionnaire.
Evaluation of physiologically-based pharmacokinetic (PBPK) models: Concentration-time profile | 24 hours
  Evaluation of the predictive performance of PBPK models by assessing whether the observed concentration-time profiles were within the 5th-95th percentile of the population prediction of the PBPK models.
Evaluation of physiologically-based pharmacokinetic (PBPK) models: M/P ratio | 24 hours
  Evaluation of the predictive performance of PBPK models by assessing whether the observed Milk-to-plasma ratio were within the 5th-95th percentile of the population prediction of the PBPK models.
Evaluation of physiologically-based pharmacokinetic (PBPK) models: Cmax | 24 hours
  Evaluation of the predictive performance of PBPK models by assessing whether the observed maximum concentration (Cmax) were within the 5th-95th percentile of the population prediction of the PBPK models.
Evaluation of physiologically-based pharmacokinetic (PBPK) models: AUC | 24 hours
  Evaluation of the predictive performance of PBPK models by assessing whether the observed Area-under-the-curve (AUC) were within the 5th-95th percentile of the population prediction of the PBPK models.
Evaluation of physiologically-based pharmacokinetic (PBPK) models: DID | 24 hours
  Evaluation of the predictive performance of PBPK models by comparing the predicted daily infant dosage (DID) with the calculated DID [The daily infant dosage (DID)(mg/d) = ∑(total drug concentration in each milk collection x expressed milk volume in each milk collection), calculated from the concentrations found in the human milk samples].
Evaluation of physiologically-based pharmacokinetic (PBPK) models: RID | 24 hours
  Evaluation of the predictive performance of PBPK models by comparing the predicted relative infant dose (RID) with the calculated RID [The relative infant dose (RID)(%) = [eDID (mg/kg/d)/Maternal Dosage (mg/kg/d)] x 100].

CONTACTS AND LOCATIONS:
Overall Officials: Anne Smits, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Del Ciampo LA, Del Ciampo IRL. Breastfeeding and the Benefits of Lactation for Women's Health. Rev Bras Ginecol Obstet. 2018 Jun;40(6):354-359. doi: 10.1055/s-0038-1657766. Epub 2018 Jul 6. PMID 29980160
- [Background] Saha MR, Ryan K, Amir LH. Postpartum women's use of medicines and breastfeeding practices: a systematic review. Int Breastfeed J. 2015 Oct 28;10:28. doi: 10.1186/s13006-015-0053-6. eCollection 2015. PMID 26516340
- [Background] Anderson PO. Drugs in Lactation. Pharm Res. 2018 Feb 6;35(3):45. doi: 10.1007/s11095-017-2287-z. PMID 29411152
- [Background] Anderson PO, Sauberan JB. Modeling drug passage into human milk. Clin Pharmacol Ther. 2016 Jul;100(1):42-52. doi: 10.1002/cpt.377. Epub 2016 May 13. PMID 27060684
- [Background] Koshimichi H, Ito K, Hisaka A, Honma M, Suzuki H. Analysis and prediction of drug transfer into human milk taking into consideration secretion and reuptake clearances across the mammary epithelia. Drug Metab Dispos. 2011 Dec;39(12):2370-80. doi: 10.1124/dmd.111.040972. Epub 2011 Sep 22. PMID 21940904
- [Background] Kimura S, Morimoto K, Okamoto H, Ueda H, Kobayashi D, Kobayashi J, Morimoto Y. Development of a human mammary epithelial cell culture model for evaluation of drug transfer into milk. Arch Pharm Res. 2006 May;29(5):424-9. doi: 10.1007/BF02968594. PMID 16756089
- [Background] McNamara PJ, Burgio D, Yoo SD. Pharmacokinetics of cimetidine during lactation: species differences in cimetidine transport into rat and rabbit milk. J Pharmacol Exp Ther. 1992 Jun;261(3):918-23. PMID 1602396
- [Background] Nauwelaerts N, Deferm N, Smits A, Bernardini C, Lammens B, Gandia P, Panchaud A, Nordeng H, Bacci ML, Forni M, Ventrella D, Van Calsteren K, DeLise A, Huys I, Bouisset-Leonard M, Allegaert K, Annaert P. A comprehensive review on non-clinical methods to study transfer of medication into breast milk - A contribution from the ConcePTION project. Biomed Pharmacother. 2021 Apr;136:111038. doi: 10.1016/j.biopha.2020.111038. Epub 2021 Jan 30. PMID 33526310
- [Background] Garessus EDG, Mielke H, Gundert-Remy U. Exposure of Infants to Isoniazid via Breast Milk After Maternal Drug Intake of Recommended Doses Is Clinically Insignificant Irrespective of Metaboliser Status. A Physiologically-Based Pharmacokinetic (PBPK) Modelling Approach to Estimate Drug Exposure of Infants via Breast-Feeding. Front Pharmacol. 2019 Jan 22;10:5. doi: 10.3389/fphar.2019.00005. eCollection 2019. PMID 30723406
- [Background] Anderson PO, Momper JD. Clinical lactation studies and the role of pharmacokinetic modeling and simulation in predicting drug exposures in breastfed infants. J Pharmacokinet Pharmacodyn. 2020 Aug;47(4):295-304. doi: 10.1007/s10928-020-09676-2. Epub 2020 Feb 7. PMID 32034606
- [Background] Maharaj AR, Edginton AN. Physiologically based pharmacokinetic modeling and simulation in pediatric drug development. CPT Pharmacometrics Syst Pharmacol. 2014 Oct 22;3(11):e150. doi: 10.1038/psp.2014.45. PMID 25353188
- [Background] Byrne JJ, Spong CY. "Is It Safe?" - The Many Unanswered Questions about Medications and Breast-Feeding. N Engl J Med. 2019 Apr 4;380(14):1296-1297. doi: 10.1056/NEJMp1817420. No abstract available. PMID 30943334
- [Background] Nauwelaerts N, Ceulemans M, Deferm N, Eerdekens A, Lammens B, Armoudjian Y, Van Calsteren K, Allegaert K, de Vries L, Annaert P, Smits A. Case Report: Bosentan and Sildenafil Exposure in Human Milk - A Contribution From the ConcePTION Project. Front Pharmacol. 2022 Jun 15;13:881084. doi: 10.3389/fphar.2022.881084. eCollection 2022. PMID 35784689
- [Background] Jones HM, Mayawala K, Poulin P. Dose selection based on physiologically based pharmacokinetic (PBPK) approaches. AAPS J. 2013 Apr;15(2):377-87. doi: 10.1208/s12248-012-9446-2. Epub 2012 Dec 27. PMID 23269526
- [Background] Mould DR, Upton RN. Basic concepts in population modeling, simulation, and model-based drug development-part 2: introduction to pharmacokinetic modeling methods. CPT Pharmacometrics Syst Pharmacol. 2013 Apr 17;2(4):e38. doi: 10.1038/psp.2013.14. No abstract available. PMID 23887688
- [Derived] Van Neste M, Nauwelaerts N, Ceulemans M, Van Calsteren K, Eerdekens A, Annaert P, Allegaert K, Smits A. Determining the exposure of maternal medicines through breastfeeding: the UmbrelLACT study protocol-a contribution from the ConcePTION project. BMJ Paediatr Open. 2024 Apr 10;8(1):e002385. doi: 10.1136/bmjpo-2023-002385. PMID 38599799
- See also: WHO Breastfeeding — https://www.who.int/health-topics/breastfeeding#tab=tab_1
- See also: FDA General Clinical Pharmacology Considerations for Neonatal Studies for Drugs and Biological Products Guidance for Industry JULY 2022 — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/general-clinical-pharmacology-considerations-neonatal-studies-drugs-and-biological-products-guidance
- See also: FDA GUIDANCE DOCUMENT Clinical Lactation Studies: Considerations for Study Design MAY 2019 — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/clinical-lactation-studies-considerations-study-design
- See also: FDA GUIDANCE DOCUMENT Physiologically Based Pharmacokinetic Analyses - Format and Content Guidance for Industry SEPTEMBER 2018 — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/physiologically-based-pharmacokinetic-analyses-format-and-content-guidance-industry
- See also: EMA Reporting of physiologically based pharmacokinetic (PBPK) modelling and simulation - Scientific guideline — https://www.ema.europa.eu/en/reporting-physiologically-based-pharmacokinetic-pbpk-modelling-simulation-scientific-guideline